CLINICAL TRIAL: NCT05260515
Title: Protecting Alzheimer Caregivers Using Technology Through Staying Sharp (PROACTS)
Brief Title: Protecting Alzheimer Caregivers Using Technology Through Staying Sharp
Acronym: PROACTS
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P30AG024978 (NIH); 5P30AG024978-18 (NIH)
Record Dates: First submitted 2022-02-07; First posted 2022-03-02 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment; Dementia Alzheimers; Old Age; Dementia; Caregiver Burden; Health Behavior; Social Behavior; Caregiver Burnout
Keywords: technology; online intervention; intervention efficacy; user experience; user adherence; remote monitoring; online platform; digital biomarker
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Caregiver Burden; Health Behavior; Social Behavior

STUDY DESIGN:
Intervention Model Description: PROACTS is a Phase I/II study to assess the efficacy of AARP Staying Sharp online health program, focusing on the health of non-professional home-based caregivers of persons with Alzheimer's disease and related dementias (ADRD). PROACTS has three aims. Aim 1 & 2 is an one-time survey study to evaluate the current uptake and utilization of Staying Sharp among caregivers. Aim 3 is a single-group intervention to assess how Staying Sharp may maintain health and function for caregivers of persons with ADRD. Participants will participate in a 4-month program with a 4-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Staying Sharp intervention (Experimental): Staying Sharp is an online intervention to promote healthy behaviors through six health pillars (Be social, Engage your brain, Manage stress, Ongoing exercise, Restorative sleep, and Eat right).
  Interventions: Behavioral: Staying Sharp intervention

INTERVENTIONS:
Behavioral: Staying Sharp intervention — In the Staying Sharp online program, participants have the opportunity to select which health pillars they are most interested in improving (Be social, Engage your brain, Manage stress, Ongoing exercise, Restorative sleep, and Eat right). After selecting the health pillars, participants can set plans and goals. There are designated activities in each health pillar for participants to complete, including watch videos, read articles, or play games. Participants will follow a step-by-step guide to achieve these goals. The website tracks the status of these goals.
  Participants will use Staying Sharp program for 4 months. Research staff will call participants to encourage participants to use the program. Right after the completion of the 4-month program, we will send out a survey to understand user experiences. We will follow participants for another 4 months. After 4 months follow-up, an exit study survey will be conducted either via videoconferences or in-person visits.

SUMMARY:
PROACTS is a Phase I/II study to assess the efficacy of AARP Staying Sharp online health program, focusing on the health of non-professional home-based caregivers of persons with Alzheimer's disease and related dementias (ADRD). PROACTS has three aims. Aim 1&2 is an one-time survey study to evaluate the current uptake and utilization of Staying Sharp among caregivers. Aim 3 is a single-group intervention to assess how Staying Sharp may maintain health and function for caregivers of persons with ADRD. Participants will participate in a 4-month program with a 4-month follow-up.

Aim 1&2: Characterize caregivers of persons with ADRD using Staying Sharp and evaluate user experiences of Staying Sharp.

Aim 3: Establish preliminary efficacy of Staying Sharp program.

DETAILED DESCRIPTION:
Significance: Approximately 16 million adults provide unpaid care to their loved ones with Alzheimer's disease and related disorders (ADRD). Among caregivers, 1 in 3 are older adults. For these caregivers, balancing their own health while caring for loved ones can be stressful, depressing, and feelings of hopelessness. This long-term distress can lead to higher risks of cardiovascular diseases, dementia, and mortality. Given the rise of incident dementia and caregiving, scalable interventions to support family caregivers are urgently needed.

Intervention: Staying Sharp is an online brain health intervention for older adults available through AARP since 2018. Over 400,000 AARP members have registered for this online intervention. This multi-component intervention includes a package of assessments, brain games, and educational videos and articles to maintain 6-pillars healthy behaviors. Independent of Staying Sharp, over 39 million have visited AARP's online caregiving resource center. The large number of visits not only shows high demand for caregiver support, but reveals the potential of Staying Sharp to reach tens of thousands of caregivers at greater risk by their role for increased morbidity and mortality.

Stage I/II user experience and efficacy study: While many users have registered for Staying Sharp, its efficacy has not been tested. Home-sensing technology is an ecologically valid way of testing the efficacy of health interventions. The Oregon Center of Aging & Technology (ORCATECH) has established a home-based, technology-agnostic, unobtrusive platform for more than 15 years. With this platform, we will assess how Staying Sharp may maintain brain health and function as indicated by a suite of digital biomarkers (e.g., physical activity, sleep, dietary behaviors). Our ultimate goal is to refine Staying Sharp by examining user experience and intervention efficacy and ultimately scale the program widely. To achieve this goal, we are collaborating with AARP. The Specific Aims of the study are to:

Aim 1: Characterize caregivers of persons with ADRD using Staying Sharp. We will send out a survey to registrants of Staying Sharp. We hypothesize that caregiver users are younger, predominantly women, with higher stress, and less social support than non-caregiver users. This aim will clarify the demographics and basic health conditions of caregivers who have been utilizing this online health intervention.

Aim 2: Evaluate user experiences of Staying Sharp. We will use the same survey in aim 1 to assess user experiences with a focus on the profile of sustainable use characteristics. We hypothesize caregiver users will spend more time on stress and exercise pillars than non-caregiver users. This aim will evaluate the engagement and uptake of Staying Sharp among dementia caregivers.

Aim 3: Establish preliminary efficacy of Staying Sharp intervention. Using unobtrusive home-sensing technologies, twenty newly-recruited caregivers of persons with ADRD will participate in a 4-month intervention with 4 months follow-up. We hypothesize that Staying Sharp will promote physical, mental, and social health for caregivers of persons with ADRD. A non-linear dose-response curve will be used to determine the pre- to post-intervention changes associated with Staying Sharp. This aim involves understanding interventions pointing toward refinement, modification, and adaptation for caregivers and pilot testing.

PROACTS uniquely takes an existing publicly available online health intervention and rapidly tests its efficacy using a home-based, unobtrusive technology platform to provide ecologically valid evidence of how this multi-component intervention may support health in caregivers of persons with ADRD. The PROACTS study will lay the groundwork for later stage (III/IV) effectiveness studies. Future grants (R01/PCORI) will bring together caregivers and health stakeholders to evaluate elements within Staying Sharp for ensuring a high-quality, high-impact, and scalable caregiver intervention.

ELIGIBILITY:
Aim 1&2 Inclusion Criteria:

* Current AARP Staying Sharp registrants
* Self-identifying as an unpaid, non-professional caregivers of persons with cognitive impairment (mild cognitive impairment to end-stage dementia)
* 18 years or older

Aim 1&2 Exclusion Criteria:

* Inability to speak English or read printed materials in English
* Conditions that would limit participation at entry to study (e.g. visual or hearing impairments prohibiting reading and discussing the survey)

Aim 3 Inclusion Criteria:

* Self-identifying as an unpaid, non-professional caregivers of persons with mild cognitive impairment (MCI) or end-stage dementia
* Have a desktop or a tablet
* Have reliable broadband internet and are email users
* Have no experiences using AARP Staying Sharp online health program
* Home is larger than a studio apartment (important for sensor data)
* 18 years or older

Aim 3 Exclusion Criteria:

* Inability to speak English or read printed materials in English
* Conditions that would limit participation at entry to study (e.g. visual or hearing impairments prohibiting reading and discussing the program and assessments)
* Any uncontrolled medical condition that is expected to preclude completion of the study, such as late stage cancers.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
User experience | Baseline
  User experiences of the Staying Sharp will be assessed using an user experience survey.
Physical activity | Change from baseline physical activity at 4 months
  Physical activity will be assessed using an Actigraphy smartwatch.
Socialization | Change from baseline socialization score at 4 months
  Socialization will be assessed using the passive infrared motion sensors installed on the front door to detect time out of the house.
Cognition | Change from baseline cognition at 4 months
  Everyday cognition will be assessed using commercial software (WorkTime; Toronto, Canada) installed on participants' desktops to collect time spent on the computers.
Caregiver Burden | Change from baseline caregiver burden at 4 months
  Caregiver burden will be assessed via a weekly online survey using the Zarit Burden Interview short form.
Sleep Health | Change from baseline sleep health at 4 months
  Sleep health will be assessed using a bed mat installed under participants' bed.
Dietary behaviors | Change from baseline dietary behaviors at 4 months
  Dietary behaviors will be assessed using an online survey modified from the Food Frequency Questionnaire (FFQ).

SECONDARY OUTCOMES:
Online engagement | Change from baseline engagement score at 4 months
  Activities engaged in the Staying Sharp will be examined (e.g., read articles, watch videos).

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kaye, MD, Study Director — Oregon Health and Science University; Chao-Yi Wu, PhD, Principal Investigator — Oregon Health and Science University

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD (without identifiable data) and all IPD that underlie results in a publication could be provided upon request.
Supporting Information: Study Protocol, ICF
Time Frame: After study results are published.
Access Criteria: Upon request